CLINICAL TRIAL: NCT06686121
Title: IMProving Mobility After revasCularizaTion in Peripheral Artery Disease: The IMPACT PAD Trial
Brief Title: Improving Mobility After Revascularization in Peripheral Artery Disease
Acronym: IMPACT PAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Rancho Research Institute (Unknown); University of Chicago (Other); Wake Forest University (Other); University of Pittsburgh Medical Center (Other); Emory University (Other); University of Arizona (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Mary McDermott, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00222333
Record Dates: First submitted 2024-11-08; First posted 2024-11-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication; Peripheral Vascular Disease; Mobility Limitation; Revascularization
Keywords: Behavior Change; Patient Reported Outcome Measures; Mobility; Revascularization; Peripheral artery disease; Intermittent claudication; 6-minute walk; Oxidative stress
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases; Mobility Limitation | interventions — Nitrates

STUDY DESIGN:
Intervention Model Description: Two x two factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) For the beetroot juice vs. placebo comparison, this will be a double blinded study where both the participant and the people collecting data will be blinded.
  For the home-based exercise, the participant and investigator will not be blinded, but the outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Home based exercise + nitrate rich beetroot juice (Experimental): This group will be participating in home based exercise and drinking nitrate rich beetroot juice for six months.
  Interventions: Behavioral: Home Based Exercise; Drug: Nitrate Rich Beetroot Juice
- Home-based exercise + placebo (Placebo Comparator): This group will be participating in home based exercise and drinking placebo beetroot juice with nitrate removed for six months.
  Interventions: Behavioral: Home Based Exercise; Drug: Placebo Beetroot Juice Without Nitrate
- Attention control + nitrate-rich beetroot juice (Experimental): This group will be participating in attention control and drinking nitrate rich beetroot juice for six months.
  Interventions: Drug: Nitrate Rich Beetroot Juice; Behavioral: Attention Control
- Attention control + placebo (Placebo Comparator): This group will be participating in attention control and drinking placebo beetroot juice with nitrate removed for six months.
  Interventions: Behavioral: Attention Control; Drug: Placebo Beetroot Juice Without Nitrate

INTERVENTIONS:
Behavioral: Home Based Exercise — This is a six month intervention where participants will walk at home for exercise with guidance from a study coach. They will attend two to four weekly meetings with the coach at the clinical site in the first 4 weeks following randomization, followed by once weekly telephone coaching calls for the remainder of the six-month intervention
  Arms: Home based exercise + nitrate rich beetroot juice; Home-based exercise + placebo
Drug: Nitrate Rich Beetroot Juice — Participants will drink one shot of nitrate rich beet-root juice twice daily for six months.
  Arms: Attention control + nitrate-rich beetroot juice; Home based exercise + nitrate rich beetroot juice
Behavioral: Attention Control — Participants will be asked to participate in weekly meetings with the coach in the attention control group for weeks 1-26. A staff member will present a topic from the National Institute on Aging "age pages" relevant to health, such as cancer screening or blood pressure treatment. Calls will last approximately 5-15 minutes and will focus on educational topics such as diabetes, healthy eating, and Medicare Part D.
  Arms: Attention control + nitrate-rich beetroot juice; Attention control + placebo
Drug: Placebo Beetroot Juice Without Nitrate — Participants will drink one shot of placebo beetroot without nitrate juice twice daily for six months.
  Arms: Attention control + placebo; Home-based exercise + placebo

SUMMARY:
Lower extremity revascularization combined with supervised exercise significantly improves walking performance compared to revascularization alone in people who have PAD without limb threatening ischemia. However, supervised exercise is inaccessible or burdensome for most PAD patients. Investigators hypothesize that home-based exercise combined with lower extremity revascularization will significantly improve walking performance compared to revascularization alone in patients with PAD undergoing revascularization for disabling PAD.

Investigators further hypothesize that inorganic nitrate, a major source of nitric oxide (NO) abundant in beetroot juice, will improve walking performance after lower extremity revascularization, compared to placebo. In preclinical models, NO inhibits inflammation, neointimal hyperplasia, thrombosis, and vascular smooth muscle cell migration at sites of revascularization. NO increases angiogenesis and perfusion, repairs skeletal muscle damaged by ischemia, and stimulates mitochondrial activity.

In a randomized clinical trial with a 2 x 2 factorial design, the trial will test the following two primary hypotheses in 386 patients randomized within three months of a successful lower extremity revascularization for disabling PAD: First, that home-based exercise combined with lower extremity revascularization will improve six-minute walk distance more than revascularization alone at 6-month follow-up (Primary Aim #1). Second, that nitrate-rich beetroot juice combined with lower extremity revascularization will improve six-minute walk, compared to placebo combined with revascularization at 6-month follow-up (Primary Aim #2).

DETAILED DESCRIPTION:
More than 300,000 surgical or endovascular lower extremity revascularization procedures are performed annually for Medicare beneficiaries who have lower extremity peripheral artery disease (PAD) without limb threatening ischemia, and rates of these procedures are increasing. In these patients, revascularization typically improves, but does not eliminate, PAD related walking impairment. Lower extremity revascularization combined with supervised exercise significantly improves walking performance compared to revascularization alone in people who have PAD without limb threatening ischemia. However, supervised exercise is inaccessible or burdensome for most PAD patients. Investigators hypothesize that home-based exercise combined with lower extremity revascularization will significantly improve walking performance compared to revascularization alone in patients with PAD undergoing revascularization for disabling PAD.

Investigators further hypothesize that inorganic nitrate, a major source of nitric oxide (NO) abundant in beetroot juice, will improve walking performance after lower extremity revascularization, compared to placebo. In preclinical models, NO inhibits inflammation, neointimal hyperplasia, thrombosis, and vascular smooth muscle cell migration at sites of revascularization. NO increases angiogenesis and perfusion, repairs skeletal muscle damaged by ischemia, and stimulates mitochondrial activity. A large body of evidence, assembled over more than 25 years, supports our hypothesis that inorganic nitrate (such as that in nitrate-rich beetroot juice) will improve walking performance and other lower extremity outcomes after lower extremity revascularization.

Effective, accessible, and safe therapies are needed to enhance the benefits and improve durability of lower extremity revascularization. Therefore, in a randomized clinical trial with a 2 x 2 factorial design, the trial will test the following two primary hypotheses in 386 patients randomized within three months of a successful lower extremity revascularization for disabling PAD: First, that home-based exercise combined with lower extremity revascularization will improve six-minute walk distance more than revascularization alone at 6-month follow-up (Primary Aim #1). Second, that nitrate-rich beetroot juice combined with lower extremity revascularization will improve six-minute walk, compared to placebo combined with revascularization at 6-month follow-up (Primary Aim #2). In Secondary Aims, the trial will establish whether home-based exercise, compared to control, and whether nitrate-rich beetroot juice, compared to placebo, improve the Walking Impairment Questionnaire and the PROMIS Mobility Questionnaire and prevent hemodynamic failure of the revascularized vessel. In exploratory aims, the trial will test the effects of the interventions on plasma nitric oxide bioavailability. If our hypotheses are correct, results of this trial will have a major impact on improving mobility in the large and growing number of people undergoing revascularization for disabling PAD.

ELIGIBILITY:
Inclusion Criteria:

Successful lower extremity revascularization for disabling PAD performed at least 30 days before baseline testing and between 30 and 100 days before randomization.

Exclusion Criteria:

1. History of leg amputation, not including toe and partial foot amputation
2. Active gangrene
3. Active limb threatening ischemia
4. Already exercising at a level consistent with exercise intervention, using investigator discretion.
5. Unstable angina
6. Unwilling to drink study beverages
7. Unwilling to adhere to the interventions and complete follow-up testing
8. Currently taking sildenafil, tadalafil, or related drugs.
9. Unwilling to accept randomization into either group (home-based exercise or attention control)
10. Currently consuming beetroot juice, oral nitrate or nitrite, or a beetroot supplement and/or unwilling to avoid beetroot juice during the study. Participants will be asked to discontinue these items for 30 days before baseline testing and throughout the clinical trial. If the potential participant is unwilling to refrain from taking these items, they will not be eligible for the clinical trial.
11. History of kidney stones that requires minimized intake of oxalate. Potential participants who need to minimize oxalate intake will be excluded from the trial.
12. Baseline blood pressure <100/45.
13. Wheelchair confinement or requiring a walker to ambulate
14. Walking is limited by a condition other than PAD
15. Current foot ulcer
16. Planned major surgery, coronary revascularization, or lower extremity revascularization during the next 12 months
17. Major medical illness including lung disease requiring oxygen, Parkinson's disease, or a life-threatening illness with life expectancy less than six months.
18. Allergy to beetroot juice
19. Currently consuming one cup or more of beets daily. Participants will be asked to decrease beet consumption to less than one cup of beets per day for 14 days before baseline testing and throughout the clinical trial. If the potential participant is unwilling to refrain from daily beet consumption of one cup or more for 30 days before the trial and during the trial, they will not be eligible for the clinical trial.
20. Participation in or completion of a clinical trial in the previous three months, using investigator discretion for trials that may not impact study participation or outcome measures of the IMPACT PAD Trial.
21. Visual impairment that limits walking ability.
22. Unable to communicate in English, unless the participant communicates in Spanish and is enrolled at a site that can deliver the intervention in Spanish. All sites with a Spanish speaking coordinator and interventionist will be able to enroll Spanish-speaking participants. While investigators aim to be as inclusive as possible, resources are not available to allow inclusion of people speaking languages that are not Spanish or English.
23. Using a mouthwash containing chlorhexidine or cetylpyridinium chloride or a mouthwash determined to be bactericidal and unwilling to discontinue.
24. Planning to begin a supervised treadmill exercise program in the next 12 months.
25. Heart attack or stroke in previous three months prior to baseline testing.
26. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2032-02-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Distance 6-month change | Baseline to 6-month follow-up
  Distance walked in six minutes

SECONDARY OUTCOMES:
Walking Impairment Questionnaire (WIQ) Distance Score 6-month change | Baseline to 6-month follow-up.
  Patient reported ability to walk long distances. Score Range 0-100, 100 is best.
Walking Impairment Questionnaire (WIQ) Distance Score 12-month change | Baseline to 12-month follow-up
  Patient reported ability to walk long distances. Score Range 0-100, 100 is best.
PROMIS Mobility Questionnaire Score 6-month change | Baseline to 6-month follow-up
  Patient report of mobility in daily living. Score range is from zero to infinity and a higher score means a better outcome.
PROMIS Mobility Questionnaire Score 12-month change | Baseline to 12-month follow-up.
  Patient report of mobility in daily living. Score range is from zero to infinity and a higher score means a better outcome.
Prevention of Hemodynamic Failure of The Revascularized Vessel | Baseline to 12 month follow-up
  Hemodynamic failure consists of loss of patency of the revascularized vessel. The outcome will be adjudicated as a categorical outcome. Medical records between randomization and final follow-up will be obtained and reviewed by the IMPACT PAD adjudication committee, consisting of field center investigators and an interventional cardiologist. Participants who meet pre-defined criteria for hemodynamic failure of the revascularized vessel.
Change in 6-minute walk distance | 12 month follow-up
  Change in 6-minute walk distance between baseline and 12-month follow-up

OTHER OUTCOMES:
Six-Minute Walk Distance | Baseline to six-month follow-up at the time point that is twenty-four hours after the final study drink
  Change in six-minute walk distance 24 hours after the final study beverage
Plasma Nitrite Levels | Baseline to 6-month follow-up
  Change in plasma nitrite levels in the blood at 6-month follow-up
BH4/BH2 6-month change | Baseline to 6-month follow-up
  Change in BH4/BH2 ratio
Progression of PAD | Baseline to 12-month follow-up
  Determine whether home-based walking exercise, compared to attention control prevents progression of PAD, defined by any new lower extremity revascularization, acute limb ischemia, or amputation of either lower extremity between baseline and 12-month follow-up.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Arizona, Tucson, Arizona
  - Rancho Research Institute, Downey, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the time the primary outcome manuscript is submitted for publication and will be available for up to 10 years.
Access Criteria: Per BioLINCC